CLINICAL TRIAL: NCT01958060
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Intravenous and Subcutaneous Doses of BI 1034020 in Healthy Male Volunteers (Partially Randomised, Single-blind, Placebo-controlled Within Dose Groups, Clinical Phase I Study)
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study of Single Escalating Doses of BI 1034020 Administered Intravenously or Subcutaneously to Male Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1312.1; 2011-004615-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-10-01; First posted 2013-10-08 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Healthy

ARMS (2):
- BI 1034020 intravenous part (Experimental): single rising doses
  Interventions: Drug: BI 1034020; Drug: Placebo to BI 1034020
- BI 1034020 subcutaneous part (Experimental): single rising doses
  Interventions: Drug: BI 1034020; Drug: Placebo to BI 1034020

INTERVENTIONS:
Drug: BI 1034020 — intravenous part
Drug: Placebo to BI 1034020 — intravenous part

SUMMARY:
Investigation of safety and tolerability of BI 1034020 in healthy male volunteers following intravenous (IV) infusion of subcutaneous (SC) injection of single doses and exploration of the pharmacokinetics and pharmacodynamics of BI 1034020 after single dosing and determination of the bioavailability of subcutaneous injections of BI 1034020

ELIGIBILITY:
Inclusion criteria:

1. Healthy males based upon a complete medical history, including a physical examination, vital signs (blood pressure, pulse rate), 12-lead electrocardiogram, and clinical laboratory tests
2. Age within the range of 18 to 40 years
3. Body mass index within the range of 18.5 and 29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion criteria:

1. Any finding in the medical examination (including blood pressure, pulse rate or electrocardiogram) deviating from normal and judged clinically relevant by the investigator. Pulse rate outside the range of 50-90 bpm or blood pressure outside the ranges of 90-140 for systolic and 50-90 mmHg for diastolic blood pressure if confirmed by repeat measurement
2. Any evidence of a clinically relevant concomitant disease.
3. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
4. Surgery of the gastrointestinal tract (except appendectomy).
5. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.
6. History of relevant orthostatic hypotension, fainting spells or blackouts.
7. Chronic or relevant acute infections.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Germany (2):
  - 1312.1.1 Boehringer Ingelheim Investigational Site, Biberach
  - 1312.1.2 Boehringer Ingelheim Investigational Site, Ingelheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was initiated at two centres. As one of the trial centres did not enrol any subjects by the time of premature termination of the trial; the trial was conducted only at one centre.
Pre-assignment Details: Partially randomised, placebo-controlled within dose groups, single-blind, single rising dose, multiple centres (dose escalation intravenous [iv] bridging to subcutaneous [sc] in parallel). 35 subjects were enrolled and 32 subjects were treated.
Groups:
- Placebo: Single dose administration of placebo to BI 1034020 through solution for intravenous (iv) infusion in the morning.
- BI 1034020 (5 mg/25 mL - iv); BI 1034020 (100 mg/25 mL - iv): Single dose administration of BI 1034020 (5 mg) diluted with 25mL solution for intravenous (iv) infusion in the morning.
- BI 1034020 (10 mg/25 mL - iv): Single dose administration of BI 1034020 (10 mg) diluted with 25mL solution for intravenous (iv) infusion in the morning.
- BI 1034020 (20 mg/25 mL - iv): Single dose administration of BI 1034020 (20 mg) diluted with 25mL solution for intravenous (iv) infusion in the morning.
- BI 1034020 (50 mg/25 mL - iv): Single dose administration of BI 1034020 (50 mg) diluted with 25mL solution for intravenous (iv) infusion in the morning.
Period: Overall Study
Arm/Group | Placebo | BI 1034020 (5 mg/25 mL - iv) | BI 1034020 (10 mg/25 mL - iv) | BI 1034020 (20 mg/25 mL - iv) | BI 1034020 (50 mg/25 mL - iv) | BI 1034020 (100 mg/25 mL - iv)
Started | 10 | 6 | 6 | 5 | 7 | 1
Completed | 8 | 6 | 6 | 5 | 6 (One subject in the 50 mg iv dose group did not receive complete dose of trial medication.) | 1 (One subject in the 100 mg iv dose group did not receive complete dose of trial medication.)
Not Completed | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Not treated | 2 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS):This subject set included all subjects who were dispensed study medication and were documented to have received 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1034020 (5 mg/25 mL - iv) | BI 1034020 (10 mg/25 mL - iv) | BI 1034020 (20 mg/25 mL - iv) | BI 1034020 (50 mg/25 mL - iv) | BI 1034020 (100 mg/25 mL - iv) | Total
Number analyzed (Participants) | 8 | 6 | 6 | 5 | 6 | 1 | 32
Age, Continuous [Mean (Standard Deviation); unit: Year] | 26.5 (4.3) | 32.5 (3.9) | 33.2 (3.4) | 31.4 (4.0) | 34.3 (4.0) | 23.0 (NA) — The data of only one patient is available and thus Standard Deviation is not calculable | 31.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 5 | 6 | 1 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug Related Adverse Events
Description: Percentage of subjects with investigator defined drug-related adverse events
Time Frame: from the first drug administration to end of trial, up to 50 days
Population: Treated Set (TS)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | BI 1034020 (5 mg/25 mL - iv) | BI 1034020 (10 mg/25 mL - iv) | BI 1034020 (20 mg/25 mL - iv) | BI 1034020 (50 mg/25 mL - iv) | BI 1034020 (100 mg/25 mL - iv)
Number analyzed (Participants) | 8 | 6 | 6 | 5 | 6 | 1
percentage of participants | 37.5 | 33.3 | 33.3 | 0.0 | 50.0 | 100.0

2. Secondary Outcome: Cmax
Description: Maximum measured concentration of BI 1034020 in plasma (Cmax).
Time Frame: 2h before study drug administration and 0.25h, 0.5h, 1h, 1.5h, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 48h, 72h, 96h, 168h, 336h, 504h, 672h, 840h and 1008h after drug administration on day 1.
Population: Pharmacokinetic Set (PKS): This subject set included all subjects in the treated set who provide at least 1 observation for at least 1 secondary Pharmacokinetic (PK) endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | BI 1034020 (5 mg/25 mL - iv) | BI 1034020 (10 mg/25 mL - iv) | BI 1034020 (20 mg/25 mL - iv) | BI 1034020 (50 mg/25 mL - iv)
Number analyzed (Participants) | 6 | 6 | 5 | 5
μg/mL | 1.50 (8.69) | 3.30 (17.6) | 6.90 (15.7) | 17.2 (11.5)
Statistical Analysis 1: Comparison: BI 1034020 (5 mg/25 mL - iv) vs BI 1034020 (10 mg/25 mL - iv) vs BI 1034020 (20 mg/25 mL - iv) vs BI 1034020 (50 mg/25 mL - iv); This was non confirmatory testing (Single dose). Dose proportionality of BI 1034020 following iv administration of single rising doses of 5 mg, 10 mg, 20 mg and 50 mg for Cmax was analysed; Test type: Superiority or Other; Slope = 1.0604, 95% CI 2-sided [0.9901 to 1.1308], Standard Error of Mean 0.0337 — Dose proportionality was explored using linear regression model (ANOVA).The perfect dose proportionality would correspond to a slope β of 1.PK endpoints on the log-transformed scale.Standard error (SE) of the mean is actually the SE of the slope

3. Secondary Outcome: AUC0-inf
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
  AUC0-inf could be assessed only in 50 mg iv dose group as terminal phase was below lower limit of quantification (BLQ) for other dose groups. Therefore dose proportionality for AUC0-inf could not be performed in this trial.
Time Frame: as for outcome 2
Population: Pharmacokinetic set (PKS):
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI 1034020 (50 mg/25 mL - iv)
Number analyzed (Participants) | 4
μg*h/mL | 314 (7.66)

4. Secondary Outcome: AUC0-tz
Description: Area under the concentration-time curve of the analyte in the plasma over the time interval from 0 to the last measurable time point of the dose (AUC0-tz ).
Time Frame: as for outcome 2
Population: Pharmacokinetic set (PKS)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI 1034020 (5 mg/25 mL - iv) | BI 1034020 (10 mg/25 mL - iv) | BI 1034020 (20 mg/25 mL - iv) | BI 1034020 (50 mg/25 mL - iv)
Number analyzed (Participants) | 6 | 6 | 5 | 5
μg*h/mL | 7.30 (9.60) | 20.1 (28.5) | 83.7 (94.4) | 242 (15.4)
Statistical Analysis 1: Comparison: BI 1034020 (5 mg/25 mL - iv) vs BI 1034020 (10 mg/25 mL - iv) vs BI 1034020 (20 mg/25 mL - iv) vs BI 1034020 (50 mg/25 mL - iv); This was non confirmatory testing (Single dose). Dose proportionality of BI 1034020 following iv administration of single rising doses of 5 mg, 10 mg, 20 mg and 50 mg for AUClast was analysed; Test type: Superiority or Other; Slope = 1.5629, 95% CI 2-sided [1.3426 to 1.7833], Standard Error of Mean 0.1056 — Dose proportionality was explored using the linear regression model.The perfect dose proportionality would correspond to a slope β of 1. PK endpoints on the log-transformed scale.Standard error of the mean is actually the standard error of the slope

ADVERSE EVENTS:
Time Frame: from the first drug administration to end of trial, up to 50 days
Arm/Group | Placebo | BI 1034020 (5 mg/25 mL - iv) | BI 1034020 (10 mg/25 mL - iv) | BI 1034020 (20 mg/25 mL - iv) | BI 1034020 (50 mg/25 mL - iv) | BI 1034020 (100 mg/25 mL - iv)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/5 | 0/6 | 1/1
Other Adverse Events (participants affected / at risk) | 6/8 | 3/6 | 4/6 | 3/5 | 5/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | BI 1034020 (5 mg/25 mL - iv) (N=6) | BI 1034020 (10 mg/25 mL - iv) (N=6) | BI 1034020 (20 mg/25 mL - iv) (N=5) | BI 1034020 (50 mg/25 mL - iv) (N=6) | BI 1034020 (100 mg/25 mL - iv) (N=1)
Anaphylactoid reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | BI 1034020 (5 mg/25 mL - iv) (N=6) | BI 1034020 (10 mg/25 mL - iv) (N=6) | BI 1034020 (20 mg/25 mL - iv) (N=5) | BI 1034020 (50 mg/25 mL - iv) (N=6) | BI 1034020 (100 mg/25 mL - iv) (N=1)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 2 | 1 | 1 | 4 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to a drug-related Serious Adverse event in the first subject of 100 mg BI 1034020 single iv dose group, the trial was prematurely terminated. No further iv dosing was performed and no planned sc dosing scheme was performed in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes